CLINICAL TRIAL: NCT01070953
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of EZETROL® in Usual Practice
Brief Title: EZETROL® Re-examination Study (MK0653-175)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0653-175; 2010_009
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EZETROL® 10 mg: Participants with Hypercholesterolemia treated with EZETROL®

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of EZETROL® through collecting the safety information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants Who Receives EZETROL® In Usual Medical Practice

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Hypercholesterolemia treated with EZETROL®
Sampling Method: Probability Sample
Enrollment: 4467 (Actual)
Dates: Start 2005-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- EZETROL® 10 mg: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily.
Period: Participants for Safety Evaluation
Arm/Group | EZETROL® 10 mg
Started | 4467
Completed | 3536
Not Completed | 931
Not completed — Violation of inclusion criteria | 612
Not completed — Off-label use | 283
Not completed — Duplicated participants | 22
Not completed — Treatment prior to date of contract | 8
Not completed — Uncontracted participants | 4
Not completed — Violation of inclusions & off label use | 1
Not completed — Duplicated participants & off-label use | 1
Period: Participants for Efficacy Evaluation
Arm/Group | EZETROL® 10 mg
Started | 3536
Completed | 3309
Not Completed | 227
Not completed — No efficacy evaluation | 119
Not completed — Lack of treatment period (<28 days) | 106
Not completed — Unknown date of efficacy evaluation | 2

BASELINE CHARACTERISTICS:
Arm/Group | EZETROL® 10 mg
Number analyzed (Participants) | 3536
Age, Customized [Number; unit: participants]
  age < 20 | 4
  20 ≤ age < 30 | 25
  30 ≤ age < 40 | 186
  40 ≤ age < 50 | 682
  50 ≤ age < 60 | 1091
  60 ≤ age < 70 | 1023
  70 ≤ age < 80 | 451
  80 ≤ age < 90 | 72
  age ≥ 90 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1861
  Male | 1675

OUTCOME MEASURES:

1. Primary Outcome: Participants With Any Clinical and/or Laboratory Adverse Experience While Being Treated With EZETROL® Within 14 Days After Treatment Discontinuation
Description: Participants who recieved EZETROL® and experienced any adverse event related or unrelated to EZETROL®, within 14 days after treatment.
Time Frame: Up to 14 days after treatment discontinuation
Measure: Number; unit: participants
Arm/Group | EZETROL® 10 mg
Number analyzed (Participants) | 4467
participants | 257

2. Primary Outcome: Mean Percent Change From Baseline to Treatment in Lipid Parameters
Description: The mean percent change from baseline to treatment in lipid parameters (total cholesterol [TC], low-density lipoprotein [LDL] cholesterol, high-density lipoprotein [HDL] cholesterol, triglycerides[TG]) in participants who received EZETROL over 4 weeks and then had available laboratory results in Lipid Parameters.
Time Frame: Baseline to 4 weeks
Population: 3,309 subjects were analyzed for the efficacy
  evaluation; 227 of the enrolled subjects did not complete the study and were excluded
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | All Participants
Number analyzed (Participants) | 3309
percentage of change
  TC (n = 2439) | -21.23 (21.16)
  HDL (n = 1928) | 3.47 (19.81)
  LDL (n = 1774) | -24.06 (33.49)
  TG ( n = 2083) | -10.37 (45.05)

3. Primary Outcome: Overall Efficacy Evaluation of EZETROL®
Description: Participants who received EZETROL over 4 weeks and then have been evaluated for overall efficacy assessment by investigator showing to be improved, unchanged or worsened.
Time Frame: Baseline to 4 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | EZETROL® 10 mg
Number analyzed (Participants) | 3309
participants
  Improved | 3029
  Unchanged | 241
  Worsened | 39
  Total | 3309

ADVERSE EVENTS:
Time Frame: Year 1 through Year 6.
Groups:
- EZETROL Year 1: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 1.
- EZETROL Year 2: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 2.
- EZETROL Year 3: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 3.
- EZETROL Year 4: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 4.
- EZETROL Year 5: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 5.
- EZETROL Year 6: Participants with Hypercholesterolemia and Homozygous Familial Hypercholesterolemia(HoFH) treated with EZETROL® 10 mg once daily in Year 6.
Arm/Group | EZETROL Year 1 | EZETROL Year 2 | EZETROL Year 3 | EZETROL Year 4 | EZETROL Year 5 | EZETROL Year 6
Serious Adverse Events (participants affected / at risk) | 0/67 | 3/1135 | 18/1039 | 9/766 | 4/154 | 2/375
Other Adverse Events (participants affected / at risk) | 0/67 | 5/1135 | 3/1039 | 0/766 | 0/154 | 29/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZETROL Year 1 (N=67) | EZETROL Year 2 (N=1135) | EZETROL Year 3 (N=1039) | EZETROL Year 4 (N=766) | EZETROL Year 5 (N=154) | EZETROL Year 6 (N=375)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC DISORDER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUROLEPTIC MALIGNANT SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
QUADRIPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGIOPATHY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZETROL Year 1 (N=67) | EZETROL Year 2 (N=1135) | EZETROL Year 3 (N=1039) | EZETROL Year 4 (N=766) | EZETROL Year 5 (N=154) | EZETROL Year 6 (N=375)
FATIGUE (General disorders) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No